CLINICAL TRIAL: NCT02753764
Title: Effects of p38 Inhibitor AZD7624 in Corticosteroid Resistant Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Donald Leung, MD, PhD, Prinicipal Investigator, National Jewish Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-2995
Record Dates: First submitted 2016-04-18; First posted 2016-04-28 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Corticosteroid Resistant (CR) Asthmatics
MeSH Terms: conditions — Asthma | interventions — AZD7624; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal control (No Intervention): Health volunteers will be recruited as an additional control group.
- Corticosteroid sensitive (CS) asthmatics (Other): After the initial visit, asthmatics will be given oral prednisone for 1 week and patients will return for the spirometer assessment. Patients will be defined as CR if <10% improvement in FEV1 % predicted is observed and as CS in >12% improvement in FEV1% predicted is observed.
  Interventions: Drug: prednisone
- Corticosteroid resistant (CR) asthmatics active (Active Comparator): The study will have a 1 week oral corticosteroid (OSC) run-in period. Subjects unresponsive to OCS will be defined as corticosteroid resistant (CR) and randomized to two crossover treatment sequences consisting of 4 weeks of inhaled AZD7624 or placebo, followed by 4 weeks of a washout period, and another 4 weeks of placebo or ASD7624
  Interventions: Drug: AZD7624; Drug: prednisone; Drug: Placebo
- Corticosteroid resistant (CR) asthmatics placebo (Placebo Comparator): The study will have a 1 week oral corticosteroid (OSC) run-in period. Subjects unresponsive to OCS will be defined as corticosteroid resistant (CR) and randomized to two crossover treatment sequences consisting of 4 weeks of inhaled AZD7624 or placebo, followed by 4 weeks of a washout period, and another 4 weeks of placebo or ASD7624
  Interventions: Drug: AZD7624; Drug: prednisone; Drug: Placebo

INTERVENTIONS:
Drug: AZD7624
  Arms: Corticosteroid resistant (CR) asthmatics active; Corticosteroid resistant (CR) asthmatics placebo
Drug: prednisone — oral prednisone 20 mg bid for one week
  Arms: Corticosteroid resistant (CR) asthmatics active; Corticosteroid resistant (CR) asthmatics placebo; Corticosteroid sensitive (CS) asthmatics
Drug: Placebo
  Arms: Corticosteroid resistant (CR) asthmatics active; Corticosteroid resistant (CR) asthmatics placebo

SUMMARY:
This is a double-blind, placebo controlled 4 week crossover study to investigate the efficacy and safety of AZD7624 (an inhaled p38 inhibitor) in corticosteroid resistant (CR) asthmatics. For the purpose of this study 10 symptomatic CR asthma patients with a FEV1% predicted <80% and normal bronchodilator response, 10 CS asthmatics and 10 healthy controls will be recruited.

DETAILED DESCRIPTION:
In Part A of the study, p38 MAPK activation will be measured in CR asthmatics and compared to CS asthmatics. Assessment of p38 MAPK activation in whole blood samples from 5 CR and 5 CS asthma patients will be performed. After fulfilling all enrollment criteria blood samples will be collected from asthma patients at Visit 1 for the whole blood evaluation of MAPK activation by flow cytometry.

After the initial visit, asthmatics will be given oral prednisone for 1 week and patients will return for the spirometry assessment. Patients will be defined as CR if <10% improvement in FEV1 % predicted is observed and as CS if >12% improvement in FEV1 % predicted is observed. If at least 2 fold increase in p-p38 MAPK expression in CD14+ cells of CR asthma patients is demonstrated when compared to CS asthmatics, Part B will be triggered. If no difference in p38 MAPK phosphorylation will be observed in monocytes of CR and CS asthmatics by flow cytometry assessment, the study will be terminated.

In Part B of the study, CR asthmatics will be randomized for treatment with AZD7624 or placebo for one month in a cross over design; the ability of AZD7624 to inhibit p38 MAPK activity will be assessed in CR patients. Five CR asthma patients from Part A may also take part in Part B. Additional CR (n=10 total patients required) and CS asthmatics (n=5) will be recruited in part B.

Baseline levels of p38 MAPK and other biomarkers will also be assessed in CR asthmatics and compared to both CS asthmatics and healthy volunteers. Patients will be enrolled and assessed for baseline p38 MAPK activation as above in peripheral blood. Patients will be re-defined as CR or CS as above based on changes in the lung function after 1 week of oral prednisone burst as above. Levels of p38 MAPK activity and other biomarkers will be compared between CR and CS patients (n=10 in each group based on recruitment for Part A and Part B) and also compared to healthy volunteers (n=10). After 1 week following oral prednisone burst, CR patients will return to undergo bronchoscopy with the collection of BAL and bronchial epithelial brushes. Blood samples will be collected for evaluation of p38 MAPK activation. CS patients will not undergo bronchoscopy, but will give a blood sample one week after oral prednisone burst for the analysis of p38 MAPK activation. Blood samples will also be collected from healthy controls during the initial visit to assess p38 MAPK activation. CR patients will be randomized for treatment with p38 inhibitor AZD7624 or placebo (5 patients per group). After 4 weeks of treatment with AZD7624 or placebo, CR patients will undergo additional bronchoscopy with the collection of BAL, brushes and blood. Patients will be monitored for adverse events during the trial. After completion of first block of cross over treatment, CR patients will undergo a 1 month wash-out period, after which, they will return for induced sputum and blood collection, and then undergo the second crossover period with AZD7624 or placebo. After the second 4 week treatment block, patients will come for sputum induction and blood collection. In CR asthma patients assessment of lung function, asthma control, airway hyperreactivity, p38 MAPK activation in peripheral blood, BAL, induced sputum samples and cellular responsiveness to corticosteroids before and after treatment with AZD7624 will be performed.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic Subjects

* Males and women of non-childbearing potential aged 18-65 of any racial or ethnic background, who are physically and mentally able to cooperate with the proposed tests and procedures and who are able to give informed consent.
* Asthma defined by symptoms and/or a doctor's diagnosis compatible with asthma as per 2014 GINA Guidelines.
* Symptomatic patients (ACQ>1.25) with FEV1 % predicted 80%, currently taking ICS or ICS/LABA. Patients should demonstrate normal bronchodilator response, i.e. there must be equal or greater than 12% or 200ml improvement in FEV1 post-bronchodilator (albuterol).
* Females must have a negative pregnancy test at Visit 1, must not be lactating and must be of non-childbearing potential, by fulfilling one of the following criteria:

  * Postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all possible exogenous hormonal treatments and luteinising hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range (at Visit 1)
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Males must be surgically sterile or agree to use an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of investigational product to prevent pregnancy in a partner.
* A weight of ≥50 kg (measured at Visit 1)

Healthy Controls

* Subjects must be 18 to 65 years old, who are physically and mentally able to cooperate with the proposed tests and procedures and who are able to give informed consent.
* They must have no respiratory or cardiac symptoms (cough, phlegm, wheeze, dyspnea) and no physician diagnosed cardiac or respiratory disease.
* No allergic history.
* FEV1≥ 80%
* Females must have a negative pregnancy test at Visit 1, must not be lactating and must be of non-childbearing potential, by fulfilling one of the following criteria:

  * Postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all possible exogenous hormonal treatments and luteinising hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range (at Visit 1)
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* A weight of ≥50 kg (measured at Visit 1)

Exclusion Criteria:

* An FEVl <60% predicted post albuterol bronchodilator.
* Oral steroid use within the past 6 weeks.
* Acute respiratory illness within 6 weeks of the study.
* Another pulmonary disease expected to affect participation in the study or the measurements to be examined.
* Pregnancy.
* Smoking in last year or prior smoking history of more than 10 pack years.
* Previous randomization to treatment in the present study (at Visit 1)
* Participation in another clinical study with any novel investigational medicine product within 3 months before the first dose of investigational product in this study (at Visit 4)
* Previously intake of any p38 inhibitor (same class as AZD7624)
* Significant disease or disorder other than asthma (e.g. cardiovascular; pulmonary as e.g. tuberculosis and cystic fibrosis; gastrointestinal, liver; neurological; musculoskeletal; endocrine; metabolic; malignant; psychiatric; major physical impairment) which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study (at Visit 1)
* Any clinically relevant abnormal findings in clinical chemistry, haematology and urinalysis, which, in the opinion of the investigator, may put the patient at risk because of participation in the study (for CR patients only at Visit 3a)
* Any clinically relevant abnormal findings in physical examination, pulse or blood pressure which, in the opinion of the investigator, may put the patient at risk because of participation in the study (at Visit 1)
* History or family history of muscle diseases (at Visit 1)
* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following (CR patients, at Visit 3a):

  * Systolic blood pressure (SBP) above 140 mmHg if <60 years of age and above 150 mmHg if ≥60 years of age
  * Diastolic blood pressure (DBP) above 90 mmHg
  * Pulse <50 or >100 bpm
* Unstable angina pectoris or stable angina pectoris classified higher than Canadian Cardiovascular Society (CSS) class 2. History of hospitalization within 12 months caused by heart failure or a diagnosis of heart failure higher than New York Heart Association (NYHA) class II. Acute myocardial infarction within 6 months of screening (CR patients, Visit 3a).
* Treatment with strong CYP3A inhibitors (like erythromycin and itraconazole), within 4 weeks prior to randomization (CVR patients, Visit 4). Patients on anticoagulation treatment.

Healthy Controls

* Evidence on history, physical examination, or screening spirometry of Lung disease or other disease that will affect participation in the study or the measurements to be examined.
* Smoking in the last year or prior smoking history of more than 10 pack years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01; Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
P38 MAPK activation (as measured by phosphorylation) in the whole blood samples by flow cytometry. | 4 months
P38 MAPK activation in the whole blood samples by flow cytometry and p38 MAPK expression in BAL and induced sputum macrophages by immunostaining and microscopy imaging before and after p38 inhibitor treatment vs placebo in CR asthma patients | 4 months
  Evaluate MAPK activation in the whole blood samples by flow cytometry and pMAPK expression in BAL and induced sputum macrophages by immunostaining and microscopy imaging before and after p38 inhibitor AZD7624 treatment vs placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided